CLINICAL TRIAL: NCT02397655
Title: Screening Carotid Artery and Intracranial Arteries by Ultrasound in Chinese Population With Transient Ischemic Attack and Ischemic Stroke: a Multi-center Registry Study
Brief Title: Vascular Ultrasound Screening in Patients With Ischemic Cerebrovascular Disease: a Multi-center Registry Study
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The First Affiliated Hospital of Shanxi Medical University (Other); Liaocheng Brains Hospital (Unknown); Tianjin Huanhu Hospital (Other); Baotou Central Hospital (Other); The First Hospital of Jilin University (Other); First Affiliated Hospital of Harbin Medical University (Other); First Hospital of China Medical University (Other); LanZhou University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The First Affiliated Hospital of Soochow University (Other); Anhui Provincial Hospital (Other Government); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); ZhuHai Hospital (Other); Fujian Provincial Hospital (Other); Mianyang Central Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Brains Hospital of Hunan Province (Unknown); Henan Provincial People's Hospital (Other); Luoyang Central Hospital (Other); National Health and Family Planning Commission Stroke Prevention Engineering Committee (Unknown); Dalian Municipal Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VUS-ICVD
Record Dates: First submitted 2015-03-18; First posted 2015-03-25 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: stroke; ischemia; atherosclerosis; ultrasonography
MeSH Terms: conditions — Stroke; Ischemia; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this multicenter study is to investigate the extra-/intra-cranial atherosclerosis distribution pattern in chinese populations with transient ischemic attack and ischemic stroke and analyze the influencing factors of atherosclerosis distribution pattern.

DETAILED DESCRIPTION:
In this multicenter study, carotid artery color doppler flow imaging and transcranial color code doppler or transcranial doppler will be used to screen the extra-/intra-cranial vessels in chinese populations with transient ischemic attack and ischemic stroke. The aim of this study is to investigate the extra-/intra-cranial atherosclerosis distribution pattern in chinese populations and analyze the influencing factors of atherosclerosis distribution pattern.

1. Ultrasound examinations procedures: According to the guidelines of vascular ultrasonography published by the Chinese Medical Doctor Association (CMDA) in 2009. The stenosis degrees of carotid artery, vertebral artery, subclavian artery as well as the middle cerebral artery are evaluated followed the criteria we published previously (references 1-4).

2. Radiology examinations procedures: Enrolled patients receive CT or MRI examinations to determine the presence and the location of cerebral infarction. If necessary, patients receive CT angiography (CTA) or MRI angiography (MRA) examinations to confirm the degrees of vessel stenosis.

3. The data collected in this study including:

1. The general informations of enrolled subjects, which include name, gender, age, resident address, telephone number.Each subject is assigned an unique identification number.
2. The history of stroke risk factors, which include 1) hypertension; 2) atrial fibrillation; 3) smoking; 4) dyslipidemia; 5) diabetes mellitus; 6) lack of physical activity (the standard of physical activity is ≥ 3 times per week and ≥30 min per time and the duration time ≥ 1 year);7) obvious overweight or obesity (BMI ≥ 26.0 Kg/m2);8) with family history of stroke.
3. The medicines used within recent 2 weeks, the surgery name (such as stenting, carotid endarterectomy)if any.
4. The results of vascular ultrasonography, ultrasonic cardiogram, radiology examinations, laboratory tests results (blood glucose, lipoproteins pattern, homocystein, C reactive protein, fibrinogen)

4. Statistic analysis plans The Statistical Package for Social Sciences (SPSS version 22.0) software was used for the statistical analyses.

1. Numerical values are shown as the mean ± standard deviation (SD). The t test or One-way ANOVA is used to compare the numerical values among different groups.
2. Chi square test is used to analyze the influencing factors on the intra-/extra-cranial atherosclerosis distribution patterns and the relationship between vessel stenosis degrees and the occurence of ischemic stroke.
3. Logistic regression is used to analyze the influencing intensity of various risk factors on atherosclerosis and ischemic events.
4. A P value <0.05 was considered statistically significant.

5. Quality assurance plans:

1. The medical centers implement the projects are the stroke prevention and treatment base hospitals awarded by National Health and Family Planning Commission, P.R. China. The medical centers have the instruments required in this study.
2. Neurologists, neurosurgeons and vascular ultrasound physicians have received standard training hosted by National Health and Family Planning Commission stroke prevention engineering committee and obtained excellent records.
3. All the centers conduct the project followed the uniform implementation plans and each center guarantee the data input in time and accurately.
4. The project has the unique database and data input in uniform format.
5. There are specific staffs to check the accuracy and completeness of data.

ELIGIBILITY:
Inclusion Criteria: Hospitalized patients with age range ≥40 years and meet one of the following two criteria.

1. Patients with transient ischemic attack in recent 3 months.
2. Patients with ischemic stroke including acute and old cerebral infarction.

Exclusion Criteria:

1. cerebral hemorrhage;
2. vessel stenosis or occlusion caused by trauma,dissection or Takayasu's arteritis；
3. Stroke patients caused by patent foramen ovale.
4. Moyamoya disease;
5. Multiple sclerosis;
6. Mitochondrial myopathy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In hospital patients with transient ischemic attack and ischemic stroke.
Sampling Method: Probability Sample
Enrollment: 12012 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Hua, MD, Principal Investigator — No.45, Changchun Road, Xicheng District, Beijing, China 100053
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hua Y, Jia L, Li L, Ling C, Miao Z, Jiao L. Evaluation of severe subclavian artery stenosis by color Doppler flow imaging. Ultrasound Med Biol. 2011 Mar;37(3):358-63. doi: 10.1016/j.ultrasmedbio.2010.12.003. Epub 2011 Jan 26. PMID 21276651
- [Background] Hua Y, Meng XF, Jia LY, Ling C, Miao ZR, Ling F, Liu JB. Color Doppler imaging evaluation of proximal vertebral artery stenosis. AJR Am J Roentgenol. 2009 Nov;193(5):1434-8. doi: 10.2214/AJR.09.2624. PMID 19843764
- [Background] Hua Y, Liu BB, Ling C, Duan C, Liu Q, Miao ZR, Li SM, Ling F. Accurate assesment of the diagnosis between 50-69% and 70-99% carotid stenoses with ultrasonography. Chinese Journal of Cerebrovascular Diseases. 3(5): 211-218,2006.
- [Background] Meng XF, Hua Y, Liu BB, Ling C, Miao ZR, Jiao LQ. The diagnostic accuracy of transcranial doppler ultrasonogrphy for middle cerebral artery stenosis. Chinese Journal of Cerebrovascular Diseases. 7(6): 284-289, 2010.
- [Derived] Liu R, Gao M, Zhao X. Evaluation of collateral circulation in patients with internal carotid artery occlusion: A clinical and ultrasonographic multicenter study. Vasc Med. 2024 Dec;29(6):707-715. doi: 10.1177/1358863X241264759. Epub 2024 Sep 8. PMID 39245861

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: This cross sectional study was totally enrolled 12012 cases. After excluded 1301 cases whose basic clinical information and/or ultrasound examination data not completed, a total of 10711 cases were entered into the final statistical analysis.
Period: Overall Study
Arm/Group | Overall Study
Started | 12012
Completed | 10711
Not Completed | 1301
Not completed — data not completed | 1301

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 10711
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3628
  Male | 7083
Region of Enrollment [Number; unit: participants]
  China | 10711

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Carotid Artery or Intracranial Artery Atherosclerosis Confirmed by Vascular Ultrasonography
Description: By using color doppler ultrasonography, the common carotid after, internal carotid artery, vertebral artery and subclavian artery stenosis were examined and the stenosis degree of these arteries were evaluated and categorized as no stenosis, <50% stenosis, 50-69% stenosis 70-99% stenosis and occlusion.
  By using transcranial color-coded sonography (TCCS) and/or transcranial doppler, the middle cerebral artery, the V4 segment of vertebral artery and basilar artery were examined and the stenosis degree of these arteries were evaluated and categorized as no stenosis, mild stenosis, medium stenosis , severe stenosis and occlusion.
  Patients with one of the above arteries having >50% stenosis or occlusion evaluated by ultrasound were underwent CTA, MRA or DSA to confirmed the stenosis degree.
Time Frame: 30 days after subjects recruitment
Population: We provide the vessel numbers with its stenosis degree ≥50% stenosis (including occlusion).
Measure: Number; unit: artery numbers
Arm/Group | Overall Study
Number analyzed (Participants) | 10711
artery numbers
  common carotid artery ≥50% stenosis | 96
  internal carotid artery ≥50% stenosis | 1063
  excranial vertebral artery ≥50% stenosis | 826
  subclavian artery ≥50% stenosis | 241
  middle cerebral artery ≥50% stenosis | 1810
  intracranial segment of vertebral artery stenosis | 777
  basilar artery ≥50% stenosis | 324

ADVERSE EVENTS:
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/12012
Other Adverse Events (participants affected / at risk) | 0/12012

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less